CLINICAL TRIAL: NCT01476527
Title: Deep Brain Stimulation for the Treatment of Refractory Bipolar Disorder: Pilot Trial
Brief Title: Deep Brain Stimulation for the Treatment of Refractory Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Andres M. Lozano, Neurosurgeon, Professor of Surgery, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0696-A
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deep Brain Stimulation (Experimental): Deep Brain Stimulation (DBS) is a neurosurgical procedure involving the implantation of deep brain electrodes, connected via a subcutaneous extension wire, to an implantable pulse generator (IPG, or 'battery') that is implanted below the collarbone
  Interventions: Procedure: Deep Brain Stimulation

INTERVENTIONS:
Procedure: Deep Brain Stimulation — Deep Brain Stimulation (DBS) is a neurosurgical procedure involving the implantation of deep brain electrodes, connected via a subcutaneous extension wire, to an implantable pulse generator (IPG, or 'battery') that is implanted below the collarbone

SUMMARY:
Bipolar Disorder (BD) is among the most comon and challenging conditions in psychiatry. Although episodes of mania and hypomania define the different types of the disorder, the clinical picture is one dominated by depressed mood and agitation. The mainstay of BD treatment has thus far been pharmacologic, but many patients remain severely disabled by their condition, despite the best available medical treatment. The successful use of deep brain stimulation (DBS) in movement disorders, and its promising results in major depressive disorder (MDD), has led researchers to consider its use in highly selected refractory cases of BD. Evidence form the imaging and circuitry literature suggests that similar underlying dyfunctional anatomic structures subserve both MDD and BD, indicating that modulation of key structures, can lead to an amelioration of symptoms and mood stabilization. Here, we propose a phase I clinical trial to evaluate the safety of DBS in BD.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a complex and disabling disorder that is among the most challenging diagnoses in psychiatry. Although episodes of mania and hypomania define the different types of the disorder, the clinical picture is one dominated by depressed mood and agitation. Detection and diagnosis of BD remains a challenge, as most individuals with BD spend many years misdiagnosed as major depression disorder (MDD), often leading to under-treatment or inappropriate treatment. Several studies have attempted to elucidate features of a major depressive episode that indicate an underlying diagnosis of MDD versus bipolar depression.

During the last fifteen years, there have been significant advances in our understanding of the pathophysiology and relevant neuroanatomy and neurocircuitry underlying mood disorders. Much of that progress has been made as a result of technological advances in neuroimaging, both structural and functional.

Deep Brain Stimulation is a neurosurgical tool has been used for over twenty-five years to treat various neurologic and psychiatric conditions. DBS is believed to work by using small amounts of electricity to disrupt the activity of brain structures that produce troublesome symptoms. In the case of Parkinson's disease, DBS is successful in treating the tremor and general slowing that are major parts of that condition. DBS has also been used in psychiatric patients, both as part of treatment, in cases of Obsessive-Compulsive Disorder (OCD), and research, in cases of Depression. The successful use of deep brain stimulation (DBS) in movement disorders, and its promising results in major depressive disorder (MDD), has led researchers to consider its use in highly selected refractory cases of BD. Evidence form the imaging and circuitry literature suggests that similar underlying dysfunctional anatomic structures subserve both MDD and BD, indicating that modulation of key structures, can lead to an amelioration of symptoms and mood stabilization.

Our primary objective is to establish the safety of deep brain stimulation in a patient population with treatment refractory bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients between the age of 30-60
* DSM IV-TR diagnosis of Bipolar Disorder I or II
* Diagnosis for >12 months with a HRSD-17 score of at least 20
* Failure of medical therapy, defined as follows:

  a. Failure of a minimum of two (2) first line as well as two (2) second line treatments for bipolar mania and depression
* No neurological disease
* No other active Axis I or Axis II co-morbidity that is the focus of clinical attention, as defined by the Mini International Neuropsychiatric Interview (MINI)
* No substance abuse or substance use disorder for minimum of three months prior to study
* Able to give informed consent
* Able to comply with all testing and follow-up visit requirements defined by the Study Protocol
* Mini mental status examination (MMSE) score >25
* Pre-menopausal women must agree to use acceptable methods of birth control (radiation risk of PET)

Exclusion Criteria:

* History of psychosis, or psychotic episodes
* Alcohol or substance dependence or abuse within 6 months, excluding nicotine or caffeine.
* Current suicidal ideation, plan or intent for self-harm.
* A suicide attempt in the past 1 year
* Major medical illness, cardiac pacemaker/defibrillator, and other implanted stimulator
* Likely to relocate or move to a location distant from the study site within one year of enrollment
* Any contraindication to MRI or PET scanning

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | Change from baseline in depression scores at 3 months, 6 months and 12 months
  Hamilton Depression Rating Scale (HAMD), Montgomery-Åsberg Depression Rating Scale (MADRS)

SECONDARY OUTCOMES:
Young Mania Rating Scale | Change from baseline in manic, hypomanic scores at 3 months, 6 months and 12 months
  Significant improvement in Young Mania Rating Scale (YMRS)
Questionnaires-Quality of Life | Change from baseline in quality of life scores at 3 months, 6 months and 12 months
  Short Form Health Survey (SF36)

CONTACTS AND LOCATIONS:
Overall Officials: Andres M Lozano, MD PhD, Principal Investigator — University Health Network, Toronto; Roger McIntyre, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada